CLINICAL TRIAL: NCT05459649
Title: A Multicenter Randomized Trial of First Line Treatment for Newly Diagnosed Immune Thrombocytopenia: Standard Steroid Treatment Versus Combined Steroid and Cyclosporin
Brief Title: Combined Steroid and Cyclosporin as First-line Treatment in Adults With Primary Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSA-ITP
Record Dates: First submitted 2022-07-10; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Prednisone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclosporin plus Steroid (Experimental): Cyclosporin: started orally 1 mg/kg/d in two divided doses for 1 week, increased to 1.5 mg/kg/d for 1week, further increased to 2.5 mg/kg/d and then continued for 24 weeks. After 26 weeks of cyclosporin treatment, the dose for patients who achieved complete response was reduced by 25 mg/d every 2 weeks to ensure continuing the lowest dose that achieved the targeted serum level of cyclosporin and a safe platelet count.
  Standard regimen of steroid for a total of 10 weeks: 1 mg per kilogram of body weight for 2 weeks followed by 40 mg daily for 2 weeks, 20 mg daily for 2 weeks, 10 mg daily for 2 weeks, 5 mg daily for 1 week and 5 mg every other day for the final week.
  Interventions: Drug: Cyclosporine Oral Product; Drug: Prednisone
- Standard steroid (Active Comparator): Standard regimen for a total of 10 weeks: 1 mg per kilogram of body weight for 2 weeks followed by 40 mg daily for 2 weeks, 20 mg daily for 2 weeks, 10 mg daily for 2 weeks, 5 mg daily for 1 week and 5 mg every other day for the final week.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Cyclosporine Oral Product — A combination of cyclosporin with standard steroid in newly diagnosed ITP patients: cyclosporin was started orally 1 mg/kg/d in two divided doses for 1 week, increased to 1.5 mg/kg/d for 1week, further increased to 2.5 mg/kg/d and then continued for 24 weeks. The therapeutic serum level of cyclosporin was 75 to 150 ug/L. After 26 weeks of cyclosporin treatment, the dose for patients who achieved complete response was reduced by 25 mg/d every 2 weeks to ensure continuing the lowest dose that achieved the targeted serum level of cyclosporin and a safe platelet count; standard steroid regimen included orally prednisone for a total of 10 weeks: 1 mg per kilogram of body weight for 2 weeks followed by 40 mg daily for 2 weeks, 20 mg daily for 2 weeks, 10 mg daily for 2 weeks, 5 mg daily for 1 week and 5 mg every other day for the final week.
  Other Names: Prednisone
  Arms: Cyclosporin plus Steroid
Drug: Prednisone — Standard steroid in newly diagnosed ITP patients: orally prednisone for a total of 10 weeks: 1 mg per kilogram of body weight for 2 weeks followed by 40 mg daily for 2 weeks, 20 mg daily for 2 weeks, 10 mg daily for 2 weeks, 5 mg daily for 1 week and 5 mg every other day for the final week.

SUMMARY:
Randomized, open-label, multicenter study to compare the efficacy and safety of cyclosporin plus standard steroid compared to standard steroid monotherapy for the first-line treatment of adults with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of 253 adults with ITP in China. Patients were randomized to cyclosporin plus standard steroid compared to standard steroid monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Newly-diagnosed, treatment-naive primary ITP;
2. Platelet counts <30×10^9/L;
3. Platelet counts < 50×10^9/L and significant bleeding symptoms (WHO bleeding scale 2 or above);
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Secondary ITP (have a known diagnosis of connective tissue diseases, malignancy, active infection, HIV infections or hepatitis B virus or hepatitis C virus infections);
3. Received first-line and second-line ITP specific treatments (e.g., steroids, intravenous immunoglobulin, TPO-RAs, rhTPO, rituximab, etc);
4. Received drugs affecting the platelet counts within 6 months before the screening visit (e.g., chemotherapy, anticoagulants, etc);
5. Severe medical condition (lung, heart, hepatic or renal disorder);
6. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Estimated)
Dates: Start 2022-07-20 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | From date of randomization until 2 years or the end of follow-up
  Nonresponse or loss of response for those who had achieved overall response (assessed in a time-to-event analysis). Overall response was defined as platelet count ≥ 30,000 per cubic millimeter and at least 2-fold increase of the baseline count and absence of bleeding.

SECONDARY OUTCOMES:
Number of patients with side effects | From date of randomization until 2 years or the end of follow-up
  Number of patients with Medication adverse events.
Number of patients with bleeding | From date of randomization until 2 years or the end of follow-up
  Number of patients with bleeding complication (WHO bleeding score)
Sustained response | From date of randomization until 2 years or the end of follow-up
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.
Overall response (OR) | From date of randomization until 2 years or the end of follow-up
  Platelet count ≥ 30,000 per cubic millimeter and at least 2-fold increase of the baseline count and absence of bleeding.
Complete response (CR) | From date of randomization until 2 years or the end of follow-up
  Platelet count > 100,000 per cubic millimeter and absence of bleeding.
Time to response | From date of randomization until 2 years or the end of follow-up
  The time from starting treatment to time of achievement of CR or OR
Duration of response | From date of randomization until 2 years or the end of follow-up
  time from OR until loss of response or until the last follow-up visit
Remission | at 12-month follow-up
  a durable platelet count ≥30×10^9/L without bleeding up to 12 months from randomization.
Rescue therapy | From date of randomization until 2 years or the end of follow-up
  any new medical intervention taken to increase the platelet count or prevent bleeding events or an increase in the dose of concomitant treatments
Associated factors of treatment failure, OR, SR and remission | From date of randomization until 2 years or the end of follow-up
  Factors that are associated with treatment failure, OR, SR and remission

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China